CLINICAL TRIAL: NCT00872456
Title: The ADHOC Project: Associations Between Diabetes Care and Haptoglobin Genotype On outComes
Brief Title: Associations Between Diabetes Care and Haptoglobin Genotype On outComes
Acronym: ADHOC
Status: Completed | Type: Observational
Sponsor: Clalit Health Services (Other)
Responsible Party: Principal Investigator, Uzi Milman, Principal Investigator, Clalit Health Services
Other Study IDs: CMC 08-0090CTIL
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Diabetes; Cardiovascular Disease; Myocardial Infarction; Stroke
Keywords: Diabetes Mellitus; Cardiovascular Disease; Haptoglobin
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases; Myocardial Infarction; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The ADHOC Cohort comprised 3044 DM individuals, treated in 47 CHS primary care clinics, that underwent haptoglobin genotyping between 2 march, 2005 and 26 September 2006. Individuals were eligible for inclusion if they had DM and were 55 years of age or older. All treatment decisions, regarding all aspects of care and follow-up of the study participants, remained at the discretion of the individual's primary care physician, who was blinded to the individual's Hp type. Hp distribution was: Hp 1-1 285 (9.4%); Hp 2-1 1248 (41.0%); Hp 2-2 1511 (49.6%).

Hypothesis: strict glucose control (HbA1c<7%) reduces the rate of cardiovascular events only to diabetic patients with the Hp 2-2 phenotype. We also postulated that, since Hp 2-2 DM individuals are at an increased genetic susceptibility for cardiovascular disease (CVD), this unique cohort merits an investigation on the associations between various CVD risk variables and CVD events and establish whether any evident association was dependent of the individual's Hp type.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients
* 55 years old or older at the time of ICARE initiation.
* Known haptoglobin genotype
* Signed informed consent for ICARE study and registry

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recruited from primary care clinics. All are diabetic patients 55 years old or older at the time of ICARE initiation (2005).
Sampling Method: Probability Sample
Enrollment: 3054 (Actual)
Dates: Start 2005-03; Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Composite of major CVD events (non fatal MI, Stroke and CVD death) | Data retrived continuously till end of 2015
  Clinical data (eg. BP, weight, smoking, etc) medications use, Lab tests and reports on CVD events will be centrally collected from patient's records and Hospital admission summaries. Admission summaries are retrieved using the computerized systems of Clalit Health Services assuring that whenever a patient in the registry is hospitalized the admission summary is retrieve. An events adjudication committee will assess each event in a blinded fashion to determine the nature of the events.

SECONDARY OUTCOMES:
Non cardiovascular death | Data retrived continuously till end of 2015
  Clinical data (eg. BP, weight, smoking, etc) medications use, Lab tests and reports on CVD events will be centrally collected from patient's records and Hospital admission summaries. Admission summaries are retrieved using the computerized systems of Clalit Health Services assuring that whenever a patient in the registry is hospitalized the admission summary is retrieve. An events adjudication committee will assess each event in a blinded fashion to determine the nature of the events.
Revascularization procedures | Data retrived continuously till end of 2015
  Clinical data (eg. BP, weight, smoking, etc) medications use, Lab tests and reports on CVD events will be centrally collected from patient's records and Hospital admission summaries. Admission summaries are retrieved using the computerized systems of Clalit Health Services assuring that whenever a patient in the registry is hospitalized the admission summary is retrieve. An events adjudication committee will assess each event in a blinded fashion to determine the nature of the events.

CONTACTS AND LOCATIONS:
Overall Officials: Uzi Milman, MD, Principal Investigator — Clalit Health Services, Haifa and Western Galilee District, Haifa, Israel.; Chen Shapira, MD, Principal Investigator — Carmel Medical Center, Clalit Health Services